CLINICAL TRIAL: NCT07402954
Title: Feasibility and Safety of Endovascular Bipolar Stimulation of the Middle Meningeal Artery for Refractory Headaches (MMA-Stim)
Brief Title: Middle Meningeal Artery Stimulation
Acronym: MMA-Stim
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-0282
Record Dates: First submitted 2026-01-26; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Migraine
Keywords: Migraine; Middle Meningeal Artery; Cadwell Cascade 32 PRO; Cadwell Guardian IONM System; Endovascular Stimulation
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single intervention arm (Experimental): Participants will undergo the planned standard-of-care middle meningeal artery (MMA) lidocaine infusion procedure. Before the lidocaine infusion begins, brief investigational electrical stimulation will be delivered using the Cadwell Cascade 32 PRO device through microwires already positioned in the artery. Stimulation will occur on each side for approximately 5 minutes per side.
  During stimulation, clinicians will record vital signs, neurologic status, and headache severity using a 0-10 scale. Continuous intra-procedural monitoring will also be performed using the Cadwell Guardian IONM System, which is FDA-approved for monitoring use.
  After stimulation is completed, participants will receive the standard MMA lidocaine infusion (50 mg over 15 minutes) as planned.
  Interventions: Device: Cadwell Cascade 32 PRO; Device: Cadwell Guardian IONM System

INTERVENTIONS:
Device: Cadwell Cascade 32 PRO — Cascade 32 PRO will be used in a way that is not part of its usual approved purpose (this is called "off-label" use) to gently deliver electrical pulses through a microcatheter.
Device: Cadwell Guardian IONM System — The Cadwell Guardian IONM System device will also be used for continuous monitoring during stimulation. The use of this device for monitoring is approved by the FDA.

SUMMARY:
This study is testing a new way to help with migraine headaches. Researchers want to see if it's safe and doable to stimulate a blood vessel in the head (called the middle meningeal artery) with microcatheters and microwires. This has never been done before for migraines and is an investigational treatment that is not part of standard migraine treatment. This stimulation would happen just before giving the standard lidocaine treatment, which is already routinely used for migraines. The goal is to see whether this new step could help improve headache outcomes.

Two FDA-cleared medical devices will be used, the Cadwell Cascade 32 PRO and the Cadwell Guardian IONM System, to perform the stimulation and monitoring. In this study, the Cascade 32 PRO will be used in a way that is not part of its usual approved purpose (this is called "off-label" use) to gently deliver electrical pulses through a microcatheter. The Cadwell Guardian IONM System will be used in its normal, FDAapproved way for continuous monitoring during stimulation.

DETAILED DESCRIPTION:
Once the patient agree to participate in this study and sign the consent form, will be asked to complete the following tests and procedures:

* Be prepped to undergo the planned standard of care MMA lidocaine infusion procedure.
* Before infusion, the doctors will briefly deliver electrical stimulation using the Cadwell Cascade 32 PRO device through microwires already in the artery. The use of this device for stimulation in the MMA is not approved by the FDA and is investigational.
* Stimulation will be given for about 5 minutes on each side.
* During stimulation with Cadwell Cascade 32 PRO, your vital signs, neurologic status, and headache severity (on a 0-10 scale) will be recorded. The Cadwell Guardian IONM System device will also be used for continuous monitoring during stimulation. The use of this device for monitoring is approved by the FDA.
* After stimulation, you will receive lidocaine infusion into the MMA (50 mg over 15 minutes) as planned.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Chronic migraine or status migrainosus, or craniofacial pain refractory to maximal medical therapy who are undergoing MMA IA lidocaine infusion.
* Subject has provided informed consent.

Exclusion Criteria:

* Known allergies to lidocaine
* Seizure disorder, history of seizures, or increased seizure susceptibility
* Intracranial vascular malformations or dural AVF
* Hemodynamic instability, any condition where brief hemodynamic shifts may pose risk
* Previous MMA intervention or craniotomy that could result in MMA occlusion
* Any implanted electronic device (pacemaker, ICD, DBS, VNS, cochlear implant, spinal cord stimulator)
* Significant cardiovascular disease (unstable angina, severe arrhythmias, recent MI)
* Severe autonomic dysfunction
* Active systemic infection
* Vulnerable populations (i.e. pregnant individuals, children, prisoners, individuals lacking decision-making capacity, persons with cognitive impairment, those unable to provide informed consent)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Safety of Bipolar Middle Meningeal Artery (MMA) Stimulation | Measured Perioperative/Periprocedural and through the immediate post-procedural period (up to 24 hours).
  Safety will be evaluated based on the ability to complete the stimulation procedure without technical failure, serious complications, or procedure-related neurological deficits.
Feasibility of Bipolar Middle Meningeal Artery (MMA) Stimulation | Measured Perioperative/Periprocedural and through the immediate post-procedural period (up to 24 hours).
  Feasibility will be demonstrated if stimulation can be successfully initiated and completed using the intended bipolar approach.

SECONDARY OUTCOMES:
Headache Severity Measured by the Visual Analog Scale (VAS) | At baseline, Perioperative/Periprocedural, immediately post-procedure, and at following post-op times 2-4 hours, 7 days, 30 days, and 90 days.
  Headache severity will be assessed using the Visual Analog Scale (VAS), a validated 0-10 cm scale in which participants indicate headache intensity by marking a point along a continuous line representing "no pain" to "worst pain."
Physiologic Responses During Stimulation | Perioperative/Periprocedural
  Physiologic responses, including heart rate, blood pressure, respiratory rate, and oxygen saturation, will be recorded during active stimulation to assess acute physiologic effects.
Patient-Reported Qualitative Outcomes | At 24 hours, 7 days, 30 days, and 90 days after the procedure.
  Patient-reported qualitative outcomes includes perceived headache relief, tolerability of the intervention, and the presence of any new or worsening symptoms.
Number of Adverse Events | Perioperative/Periprocedural, and at follow-up at 7 days, 30 days, and 90 days.
  Adverse events and serious adverse events including seizures, vascular complications, and signs of lidocaine toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kan, MD,MPH, Principal Investigator — University of Texas Medial Branch
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No